CLINICAL TRIAL: NCT04441723
Title: Comparison of Dynamic Versus Static Lag Screw Modes for Cephalomedullary Nails Used to Fix Peritrochanteric Fragility Fractures
Brief Title: Comparison of Dynamic Versus Static Lag Screw Modes for Cephalomedullary Nails Used to Fix Intertrochanteric Fragility Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Traumatologico Dr. Teodoro Gebauer Weisser (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STVSDY
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Intertrochanteric fractures; Cephalomedullary Nails; Cut-out; Cut through
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- lag screw with dynamic mode (Active Comparator): Device: Gamma 3 nail whit lag screw on dynamic mode Surgical stabilization of intertrochanteric hip fractures using two different lag screw modes
  Interventions: Device: Osteosynthesis with Gamma 3 nail , using a dynamic lag screw as a proximal fixation.
- lag screw with static mode (Active Comparator): Device: Gamma 3 nail whit lag screw on dynamic mode Surgical stabilization of intertrochanteric hip fractures using two different lag screw modes
  Interventions: Device: Osteosynthesis with Gamma 3 nail , using a static lag screw as a proximal fixation.

INTERVENTIONS:
Device: Osteosynthesis with Gamma 3 nail , using a dynamic lag screw as a proximal fixation. — Closed reduction and surgical stabilization of intertrochanteric hip fractures using Gamma 3 nail , with dynamic lag screw as proximal fixation
  Arms: lag screw with dynamic mode
Device: Osteosynthesis with Gamma 3 nail , using a static lag screw as a proximal fixation. — Closed reduction and surgical stabilization of intertrochanteric hip fractures using Gamma 3 nail , with static lag screw as proximal fixation
  Arms: lag screw with static mode

SUMMARY:
The objective of this study is to compare the failure rate between two modes of fixing the lag screw of the cephalomedullary nail.

The sample studied will be patients who have been diagnosed with a fragility intertrochanteric fracture.

Investigators hypothesis is that the dynamic mode will have a lower failure rate compared to the static mode.

DETAILED DESCRIPTION:
Intertrochanteric fragility fractures are one of the most frequent fractures in the elderly . They produce great disability and complications in our patients and they are recognized worldwide as a major public health problem.

The treatment that presents the best results is surgical treatment, since it reduces the mortality of the patients and allows early loading . Thus, avoids secondary complications to the prostration state such as pneumonia, bedsores, pulmonary embolisms, among others.

Currently, the treatment that has shown the best clinical and biomechanical results is osteosynthesis with a cephalomedullary nail, which despite having good results is not free from complications such as implant failure, loss of femoral offset.

Changes are constantly made in the design and surgical techniques of these implants in order to decrease the rate of complications.

This study will particularly assess whether there is any difference in the complication rate between dynamic versus static lag screw modes.

Biomechanical studies that compare these two lag screw modes show that axial and lateral stiffness of the femur-nail construction is greater in static mode than in dynamic modes and the torsional stiffness is greater in dynamic mode than in static modes.

There are no studies comparing the clinical results of these two variants.

ELIGIBILITY:
Inclusion Criteria:

* Low Energy Mechanism
* Hip fracture classified as 31.A1.2 - 31 A1.3 and 31.A2 in the AO classification (year 2018)

Exclusion Criteria:

* A fracture due to malignancy
* Previous contralateral fracture
* Inability to walk before the fracture
* An inability to comply with rehabilitation
* Follow-up of less than 6 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Implant failure | 6 months
  Rate of cut out , cut through.

SECONDARY OUTCOMES:
Complications | 3 weeks, 3 months , 6 months
  Rate of Infection and Non Union.
Offset | 6 months
  Changes in femoral offset

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Traumatologico, Santiago, Chile

REFERENCES:
- [Background] Kuzyk PR, Shah S, Zdero R, Olsen M, Waddell JP, Schemitsch EH. A biomechanical comparison of static versus dynamic lag screw modes for cephalomedullary nails used to fix unstable peritrochanteric fractures. J Trauma Acute Care Surg. 2012 Feb;72(2):E65-70. doi: 10.1097/ta.0b013e3182170823. PMID 22439235
- [Background] Mahomed N, Harrington I, Kellam J, Maistrelli G, Hearn T, Vroemen J. Biomechanical analysis of the Gamma nail and sliding hip screw. Clin Orthop Relat Res. 1994 Jul;(304):280-8. PMID 8020229
- [Background] Bhandari M, Swiontkowski M. Management of Acute Hip Fracture. N Engl J Med. 2017 Nov 23;377(21):2053-2062. doi: 10.1056/NEJMcp1611090. No abstract available. PMID 29166235